CLINICAL TRIAL: NCT01484379
Title: Surgical Approach for Primary Hyperparathyroidism in the Elderly - a Prospective Study
Brief Title: Surgical Approach for Primary Hyperparathyroidism in the Elderly
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulties in Recruiting patients
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: parathyroid409-11-RMBCTIL
Record Dates: First submitted 2011-12-01; First posted 2011-12-02 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Multigland Disease in Primary Hyperparathyroidism
Keywords: Primary Hyperparathyroidism; multigland disease; neck exploration; elderly
MeSH Terms: conditions — Hyperparathyroidism, Primary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- unilateral neck exploration (Experimental): unilateral neck exploration of elderly with primary hyperparathyroidism
  Interventions: Procedure: unilateral neck exploration

INTERVENTIONS:
Procedure: unilateral neck exploration — All elderly patients with primary hyperparathyroidism suspected to have a single gland disease will have a unilateral neck exploration following the index gland identification.

SUMMARY:
Following a personal observation and a retrospective analysis of the data, the investigators hypothesise that there is increased frequency of multiple gland disease in primary hyperparathyroidism in the elderly.

This study will include patients over the age of 65, diagnosed with primary hyperaprathyroidism, referred for surgery and suspected to have a single adenoma according to preoperative imaging. Surgery will begin with a focal parathyroid exploration as suspected followed by an exploration of the other gland at the same time. Data will be analysed to determine the frequency of multigland disease in this population.

ELIGIBILITY:
Inclusion Criteria:

* patient with primary hyperparathyroidism.
* patients with an indication for surgery.
* Suspected adenoma on preop images.
* minimum age of 65.

Exclusion Criteria:

* patients younger than 65.
* cases where imaging didn't locate any adenoma.
* patients who did not consent to participate in the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-12; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Frequency of multigland disease in hyperparathyroidism in the elderly. | two years

CONTACTS AND LOCATIONS:
Overall Officials: Michal Mekel, M.D, Principal Investigator — Rambam health care campus Haifa Israel
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

REFERENCES:
- [Background] Kebebew E, Duh QY, Clark OH. Parathyroidectomy for primary hyperparathyroidism in octogenarians and nonagenarians: a plea for early surgical referral. Arch Surg. 2003 Aug;138(8):867-71. doi: 10.1001/archsurg.138.8.867. PMID 12912745
- [Background] Shin SH, Holmes H, Bao R, Jimenez C, Kee SS, Potylchansky E, Lee JE, Evans DB, Perrier ND. Outpatient minimally invasive parathyroidectomy is safe for elderly patients. J Am Coll Surg. 2009 Jun;208(6):1071-6. doi: 10.1016/j.jamcollsurg.2009.01.048. Epub 2009 Apr 17. PMID 19476894
- [Background] Uden P, Chan A, Duh QY, Siperstein A, Clark OH. Primary hyperparathyroidism in younger and older patients: symptoms and outcome of surgery. World J Surg. 1992 Jul-Aug;16(4):791-7; discussion 798. doi: 10.1007/BF02067389. PMID 1413850